CLINICAL TRIAL: NCT00375999
Title: A Phase II Study of Docetaxel and Epirubicin Combination in Patients With Advanced Gastric Cancer.
Brief Title: Docetaxel and Epirubicin in Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jae Yong Cho, Chisf of Medical oncology, Gangnam Severance Hospital, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-232
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-01

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Epirubicin

ARMS (1):
- docetaxel and epirubicin (Experimental): salvage docetaxel and epirubicin
  Interventions: Drug: Docetaxel and epirubicin

INTERVENTIONS:
Drug: Docetaxel and epirubicin
  Other Names: taxotere; pharmorubicin

SUMMARY:
1.Study rationale:There is no standard regimen for the advanced and/or metastatic gastric cancer patients who relapsed after adjuvant chemotherapy or failed to first systemic chemotherapy. 2.Primary Objectives:To evaluate overall response rate according to the Response Evaluation Criteria in Solid Tumors criteria and To investigate time to response 3.Design:single-center, Open label, Phase II study. docetaxel 75mg/m2 administered on day 1 as intravenously combined with intravenous Epirubicin 60mg/m2 given day 2 every 3 weeks. 4.Primary endpoints:

1. Efficacy:overall response rate according to the Response Evaluation Criteria in Solid Tumors criteria, time to response, duration of response, and time to treatment failure.
2. Safety-Adverse events and laboratory tests, graded according to the NCI Common Toxicity Criteria for Adverse Effects (version 3.0).

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients ≥ 18 years,
* Eastern Cooperative Oncology Group performance status below 1, with histologically confirmed as gastric adenocarcinoma with inoperable and/or metastatic disease.
* Patients must have at least one target lesion with a minimum lesion size as per the Response Evaluation Criteria in Solid Tumors criteria (at least 1 unidimensional measurable lesion ≥ 20 mm in diameter by conventional CT or MRI scan, or ≥ 10 mm in diameter by spiral CT scan).
* Creatinine clearance ≥ 60ml/min (estimated creatinine clearance must be calculated at baseline for all patients.)
* Adequate major organ function : - Hematopoietic function: white blood cell >4,000/mm3 or absolute neutrophil count > 2,000/mm3, Platelet count ≥ 100,000/mm3,- Hepatic function: Bilirubin < 1.5 X upper normal limit, aspartate aminotransferase/alanine aminotransferase levels <2.5 X upper normal limit, alkaline phosphatase < 5 x upper normal limit (except in case of bone metastasis without any liver disease) - Renal function: Creatinine <1 x upper normal limit or creatinine clearance ≥ 60ml/min.

Exclusion Criteria:

* Patients must not have previously received systemic treatment (cytotoxic chemotherapy or active/passive immunotherapy) for advanced or metastatic disease.
* Adjuvant or neo-adjuvant treatment for non-metastatic (M0) disease is allowed if completed at least 6 months prior to initiation of study treatment.
* The following laboratory values: - neutrophils ≤1.5 X 109 /L, platelet count<100 X 109 /L- serum bilirubin ≥ 1.5 X upper normal limit, aspartate aminotransferase

  , alanine aminotransferase > 2.5 X upper normal limit or > 5 X upper normal limit in the case of liver metastases- Alkaline phosphatase > 2.5 X upper normal limit or 5 X upper normal limit in the case of liver metastases or > 10 X upper normal limit in the case of bone disease.
* Prior therapy with Taxotere or Epirubicin is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Yong Cho, Principal Investigator — Yonsei University
Locations (1):
- Yongdong Severance Hospital, Seoul, South Korea

REFERENCES:
- [Result] Lim JY, Cho JY, Paik YH, Lee DK, Lee SI, Park HJ, Lee SJ, Lee KS, Yoon DS, Choi SH. Salvage chemotherapy with docetaxel and epirubicin for advanced/metastatic gastric cancer. Oncology. 2007;73(1-2):2-8. doi: 10.1159/000120027. Epub 2008 Mar 10. PMID 18332648

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Salvage Chemotherapy with Docetaxel and Epirubicin for Advanced/Metastatic Gastric Cancer
Period: Overall Study
Arm/Group | Treatment Group
Started | 34
Completed | 32
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 53 [34 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: One year
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Treatment Group
Number analyzed (Participants) | 32
month | 13.4 [7.0 to 19.8]

ADVERSE EVENTS:
Arm/Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 3/34
Other Adverse Events (participants affected / at risk) | 16/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=34)
sepsis (Infections and infestations) | 1
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=34)
neutropenia (Blood and lymphatic system disorders) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No